CLINICAL TRIAL: NCT01825109
Title: Improving the Immune Response to Rotavirus Vaccine
Brief Title: Improving Rotavirus Vaccine Immune Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: European Centre for Disease Prevention and Control, SE-171, Stockholm (Unknown); The Swedish Institute for Infectious Disease Control, SE-171 82 SOLNA (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-09070
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2009-12

CONDITIONS: Healthy Infants; Mothers
Keywords: Rotavirus; Immunogenicity; vaccine, Bangladesh
MeSH Terms: interventions — Rotavirus Vaccines; Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 6 weeks RV & normal breast feeding (Experimental): Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus vaccine with no intervention in normal breastfeeding practices before and after receiving vaccine.
  Interventions: Biological: Rotavirus Vaccine & Breastfeeding
- 6 weeks RV & delayed breastfeeding (Experimental): Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration.
  Interventions: Biological: Rotavirus Vaccine & Breastfeeding
- 14 weeks RV & Normal breastfeeding (Experimental): Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus, with no intervention in normal breastfeeding practices before and after receiving vaccine.
  Interventions: Biological: Rotavirus Vaccine & Breastfeeding
- 14 weeks RV & delayed breastfeedin (Experimental): Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration.
  Interventions: Biological: Rotavirus Vaccine & Breastfeeding

INTERVENTIONS:
Biological: Rotavirus Vaccine & Breastfeeding — Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus vaccine with no intervention in normal breastfeeding practices before and after receiving vaccine.
  Arms: 6 weeks RV & normal breast feeding
Biological: Rotavirus Vaccine & Breastfeeding — Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration.
  Arms: 6 weeks RV & delayed breastfeeding
Biological: Rotavirus Vaccine & Breastfeeding — Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus, with no intervention in normal breastfeeding practices before and after receiving vaccine.
  Arms: 14 weeks RV & Normal breastfeeding
Biological: Rotavirus Vaccine & Breastfeeding — Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration.
  Arms: 14 weeks RV & delayed breastfeedin

SUMMARY:
Rotavirus is the leading cause of severe gastroenteritis in infants and young children worldwide and is estimated to account for 600,000 deaths in children <5 years of age. However, live oral enteric vaccines (e.g. OPV, cholera vaccines, typhoid vaccine) have been less immunogenic in poor communities with high levels of malnutrition and poor sanitation. Rotavirus vaccines also appear to be less immunogenic in the setting where they are most needed. High maternal antibody (IgG) to rotavirus and breast feeding near the time of vaccination may inhibit rotavirus vaccine effectiveness. We propose a quick study to look at practical ways to improve the immunogenicity of rotavirus vaccine in our own setting in Bangladesh. The objectives are to assess if delaying Rotarix vaccination will improve the immune response to the vaccine and to assess if avoiding breastfeeding in the 45 minutes before and after vaccine administration will improve the immune response to administration of Rotarix vaccine. The study will be conducted in the urban Dhaka Mirpur Community, a setting where previous rotavirus vaccine immunogenicity studies have been successfully conducted. A total of 300 infant will be randomly assigned to one of the following groups: 1) Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus vaccine with no intervention in normal breastfeeding practices before and after receiving vaccine. 2) Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration. 3) Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus, with no intervention in normal breastfeeding practices before and after receiving vaccine. 4) Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration. Blood and stool samples will be collected from infants and breast milk from mothers. The primary outcome is to determine the sero-conversion rate of anti-rotavirus IgA in different groups of infants.

DETAILED DESCRIPTION:
The study will be conducted in a suburb of Dhaka in the area of Mirpur. Mirpur is one of the 14 Thanas of Dhaka cities with a population of about one million in an area of 59 square kilometers. Mirpur Thana of Dhaka city is divided into several sections. There are 14 sections in Mirpur Thana. The area is densely populated and located 20 minutes away from the lCDDR,B's Dhaka Hospital . The population is stable with low socioeconomic conditions. The average income in the slum areas of Mirpur is Tk.4200 (about US $ 62) per month per family. 25% of fathers and 15% of mothers have more than 5 years of formal education. The study will be conducted in section 11 and 12 of Mirpur which has a population of about 500,000. We recently conducted phase I and II of the rotavirus vaccine study in this site. Several other studies (phase II ETEC, killed cholera vaccine) are ongoing in this area. Children will be identified through active surveillance of new births in the community and the study subjects will be recruited through home visits by the locally recruited field workers.

2.2 .Design : Randomized intervention trial

Study groups:

1. Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus vaccine with no intervention in normal breastfeeding practices before and after receiving vaccine.
2. Administration of Rotarix at 6 and 10 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration.
3. Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus, with no intervention in normal breastfeeding practices before and after receiving vaccine.
4. Administration of Rotarix at 14 and 18 weeks co-administered with oral polio virus. Breastfeeding will not be permitted 45 minutes prior to vaccine administration and 45 minutes after each vaccine administration.

Samples collected:

* Blood draw at the time of first dose of Rotavirus vaccine and 4 weeks after the second dose
* Breast milk sample at 6 weeks for the mothers in study groups A and B, and at 14 weeks for mothers in study groups C and D (see below for groups).
* Stool sample prior to dose one and on day 3 and 7 after each dose to look for vaccine virus shedding

ELIGIBILITY:
Inclusion Criteria:

* male or female,
* aged 6 weeks at the time of enrollment,
* written informed consent,
* free of chronic or serious medical condition as determined by history and physical exam and plan to stay in community for at least 6 months

Exclusion Criteria:

* fever (>38 C),
* acute or chronic illness,
* use of antimicrobial drug within previous 14 days,
* hypersensitivity to any of the vaccine components (see vaccine composition),
* use of any investigational drug during previous 30 days,
* any uncorrected congenital malformation of the gastrointestinal tract,
* use of any immunosuppressing drugs during the last 14 days (likelihood is remote),
* any evidence by physical exam of immunosuppresing condition,
* administration of gamma globulin or any other blood product,
* previous intussusception or abdominal surgery.

Ages: 1 Month to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of Rotavirus Vaccine | 24 months
  Sero-conversion rate of anti-rotavirus IgA

SECONDARY OUTCOMES:
anti-rotavirus IgA | 24 months
  Geometric mean concentration of anti-rotavirus IgA Enterovirus excretion in children at the time of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Mirpur, Dhaka, Bangladesh